CLINICAL TRIAL: NCT07035340
Title: EFFECTS OF INSPIRATION MUSCLE TRAINING ON NT-PROBNP, FUNCTIONAL EXERCISE CAPACITY, DAILY LIVING EXERCISE PERFORMANCE, AND QUALITY OF LIFE IN PATIENTS UNDERGOING CARDIAC RESYNCHRONIZATION THERAPY
Brief Title: Effects of IMT on Cardiac Resynchronization Therapy
Acronym: CRT-IMT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tarsus University (Other)
Responsible Party: Principal Investigator, Nurel Ertürk, Phd,PT, Tarsus University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024/42
Record Dates: First submitted 2025-06-13; First posted 2025-06-25 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-06

CONDITIONS: Cardiac Resynchronization Therapy
Keywords: inspiratory muscle training; cardiac resynchronization therapy; exercises capacity; quality of life

STUDY DESIGN:
Masking Description: Doctor who doing ekogardiography.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- İntervention group (Experimental): inspiratory muscle training
  Interventions: Other: inspiratory muscle training
- Control group (Other): Standart care
  Interventions: Other: standart care

INTERVENTIONS:
Other: inspiratory muscle training — inspiratory muscle traning MIP%40-60
  Arms: İntervention group
Other: standart care — standart care
  Arms: Control group

SUMMARY:
Patients who are followed up in the cardiology clinic with a diagnosis of CHF, who have had a CRT implant at least 1 year ago, and who do not receive cardiac rehabilitation will be included. The aim of the study is to investigate the effects of inspiratory muscle training (IMT) on exercise capacity, respiratory muscle strength, NTproBNP and quality of life.

Groups Intervention group: Treatment with IMT Control group: Standard care Study hypothesis;

1. Does IMT have an effect on exercise capacity and quality of life in patients with CRT?
2. Does IMT have an effect on NTproBNP in patients with CRT?

ELIGIBILITY:
Inclusion Criteria:

* Patients who were followed up in the cardiology clinic with a diagnosis of CHF,
* CRT implanted at least 1 year ago,
* did not receive cardiac rehabilitation,
* 45-75 years old,
* communicate in Turkish,
* NYHA II-III

Exclusion Criteria:

* orthopedic and neurological disorders that may prevent walking,
* acute respiratory tract infection in the last month,
* NYHA I were not included in this study because they were generally not hospitalised and the problems were managed with outpatient diagnosis and treatment, and patients with class IV were not included in this study because they showed severe symptoms for medical and ethical reasons and they were not wanted to be forced with this long-lasting survey application process.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2024-05-15 (Actual); Primary Completion 2025-06-15 (Actual); Study Completion 2025-06-15 (Actual)

PRIMARY OUTCOMES:
NT-proBNP | enrollment and end of the 12 week treatment
  NT-proBNP
Exercises capacity | enrollment and end of the first week of treatment
  Exercise capacity was evaluated using the 6-minute walk test (6MWT). 6MWT was performed according to the ATS/ERS criteria.
Heart rate (Exercises capacity) | enrollment and end of the first week of treatment
  Heart rate were measured using a portable pulse oximeter (Cosmed Srl, Cosmed Spiropalm, Rome, Italy), before, after and 1 minute recovery.
Quality of Life of patients | enrollment and end of the 12 week treatment
  Qality of life was assessed using the Nottingham Health Profile (NHP) self-reported tool. The NHP questionnaire evaluates six dimensions of health (pain, energy level, sleep, physical abilities, emotional reaction and social isolation) and includes 38 items. Total NHP score ranges between 0-600 and quality of life perception is negatively associated with score received

SECONDARY OUTCOMES:
Respiratory muscle strength | enrollment and end of the first week of treatment
  Respiratory muscle strength was measured with a portable, electronic mouth pressure measuring device (Micro Medical Micro RPM, Rochester, UK). Three measurements were made to obtain the best value. There should not be more than a 10% difference between the two best-measured values. Actual MIP values and percentages of expected values according to age and gender were used in the analysis
The performance of patients' activities of daily living | at enrollment and end of the 12 week treatment
  The performance of patients' activities of daily living was assessed with the Performance Measurement of Activities of Daily Living Questionnaire-8 (PMDL-8), the Turkish validity and reliability of which was performed by Ertürk et al. The PMADL-8 questionnaire for Patients with Congestive Heart Failure assesses functional limitations in CHF patients based on the ICF model. High scores indicate severe functional limitations.

CONTACTS AND LOCATIONS:
Locations (1):
- Tarsus University, Mersin, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No